CLINICAL TRIAL: NCT06806137
Title: A Phase 3a, Observer-blind, Randomized, Controlled, Study to Evaluate the Immunogenicity and Safety of an Investigational Varicella Vaccine Compared With Varivax, When Given as a Second Dose to Healthy Children, 3 Months After the Administration of a First Dose at 12 to 15 Months of Age
Brief Title: A Study on the Immune Response and Safety of the Second Dose of an Investigational Chickenpox Vaccine When Given to Healthy Children 3 Months After a First Dose at 12 to 15 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 214002; 2024-516635-27-00 (Other: EU CT Number)
Record Dates: First submitted 2025-01-31; First posted 2025-02-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Chickenpox
Keywords: Chicken pox; Investigational varicella vaccine (VNS) Varicella; Varivax (VV); Healthy Children
MeSH Terms: conditions — Chickenpox | interventions — Measles-Mumps-Rubella Vaccine; Hepatitis A Vaccines; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant
Masking Description: Observer-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VV-VV Group (Active Comparator): Participants receive 2 doses of a VV vaccine on Day 1 and Day 91. 1 dose of measles, mumps, and rubella (MMR) vaccine, 1 dose of hepatitis A vaccine (HAV), and 1 dose of PCV (either PCV 13 or Vaxneuvance or PCV 20) on Day 1. A second dose of MMR vaccine will be co-administered to the participants in countries where a second dose of MMR is recommended at 15 to 18 months of age, as per national immunization schedule.
  Interventions: Biological: Marketed varicella vaccine; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance
- VNS-VNS Group (Experimental): Participants receive 2 doses of a VNS vaccine on Day 1 and Day 91. 1 doses of MMR vaccine, 1 dose of HAV vaccine, and 1 dose of PCV (either PCV 13, Vaxneuvance or PCV 20) on Day 1. A second dose of MMR vaccine will be co-administered to the participants in countries where second dose of MMR is recommended at 15 to 18 months of age, as per national immunization schedule.
  Interventions: Biological: Investigational varicella vaccine; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance
- VV-VNS Group (Experimental): Participants receive 1 dose of VV vaccine on Day 1, 1 dose of VNS Vaccine on Day 91. 1 doses of MMR vaccine, 1 dose of HAV, and 1 dose of PCV (either PCV 13, Vaxneuvance or PCV 20) on Day 1. A second dose of MMR vaccine will be co-administered to the participants in countries where second dose of MMR is recommended at 15 to 18 months of age, as per national immunization schedule.
  Interventions: Biological: Investigational varicella vaccine; Biological: Marketed varicella vaccine; Biological: MMR vaccine; Biological: Hepatitis A vaccine; Biological: PCV (pneumococcal conjugate vaccine) 13; Biological: PCV 20; Biological: Vaxneuvance

INTERVENTIONS:
Biological: Investigational varicella vaccine — Investigational varicella vaccine administered subcutaneously.
  Arms: VNS-VNS Group; VV-VNS Group
Biological: Marketed varicella vaccine — Marketed varicella vaccine administered subcutaneously.
  Arms: VV-VNS Group; VV-VV Group
Biological: MMR vaccine — MMR vaccine co-administered subcutaneously or intramuscularly.
Biological: Hepatitis A vaccine — Hepatitis A vaccine co-administered intramuscularly.
Biological: PCV (pneumococcal conjugate vaccine) 13 — The 13-valent pneumococcal conjugate vaccine co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.
Biological: PCV 20 — The 20-valent pneumococcal conjugate vaccine co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.
Biological: Vaxneuvance — The Vaxneuvance (15-valent pneumococcal conjugate vaccine co-administered intramuscularly. In some countries PCV will only be administered depending on the availability, country's registration status and national recommendations for pneumococcal vaccination at the time of study conduct.

SUMMARY:
The purpose of this study is to evaluate the immune response and safety of GSKs investigational varicella vaccine (VNS Vaccine) compared to an already approved varicella vaccine, Varivax (VV), when administered as second dose to healthy children. 3 months after first dose at 12 to 15 months. The study will be conducted in children who have not previously contracted varicella or received a varicella vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent(s)/Legally acceptable representative (LAR)(s), who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written or witnessed/thumb printed informed consent obtained from the participant's parent(s)/LAR(s) prior to performance of any study-specific procedure.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female between, and including, 12 to 15 months of age (i.e., from the day of 1 year birthday until the day before 16 months of age) at the time of the administration of the first study interventions.
* Only for children in countries where PCV is recommended at 12 to 15 months of age as per national immunization schedule and provided as part of the study interventions: participant who previously received the primary series of PCV in the first year of life with last dose at least 60 days prior to study entry.

Exclusion Criteria:

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity to latex.
* Major congenital defects, as assessed by the investigator.
* Recurrent history of uncontrolled neurological disorders or seizures.
* History of varicella disease.
* Active untreated tuberculosis.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study interventions during the period beginning 30 days before the first dose of study interventions (Day -29 to Day 1), or their planned use during the study period.
* Planned administration of a vaccine in the period starting 30 days before the first dose and ending 43 days after the second dose of study interventions administration (Visit 3), with the exception of inactivated influenza vaccine which may be given at any time during the study and administered at a different location than the study interventions.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

  * Up to 90 days prior to the study intervention administration:

    i) For corticosteroids, this will mean prednisone equivalent >=0.5 mg/kg/day with maximum of 20 mg/day for pediatric participants. Inhaled and topical steroids are allowed.

ii) Administration of immunoglobulins and/or any blood products or plasma derivatives.

* Up to 180 days prior to study interventions administration: long acting immune-modifying drugs including among others immunotherapy (e.g., tumor necrosis factor-inhibitors), monoclonal antibodies (except the ones not interfering with the immune response to the study vaccinese.g., nirsevimab), antitumoral medication.
* Previous vaccination against measles, mumps, and rubella.
* Previous vaccination against hepatitis A virus.
* Previous vaccination against varicella virus.
* Only for children in countries where PCV is recommended at 12 to 15 months of age as per national immunization schedule and provided as part of the study interventions, participant who previously received a booster dose of any PCV.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).
* Child in care.
* Any study personnel's immediate dependents, family, or household members.
* Participants with the following high-risk individuals in their household:

  i) Immunocompromised individuals. ii) Pregnant women without documented history of varicella. iii) Newborn infants of mothers without documented history of varicella. iv) Newborn infants born less than (<) 28 weeks of gestation.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with seroresponse to Varicella Zoster Virus (VZV) anti- glycoprotein E (gE) IgG for 2 doses of VNS vaccine compared to 2 doses of VV | At Day 133 (43 days post-dose 2)
  Seroresponse is defined as post-vaccination (Day 43 post Dose 2) anti VZV gE Immunoglobulin (IgG) concentration greater than equal to (>=) 300 milli-international units per milliliter (mIU/mL).
Geometric Mean Concentration (GMC) of anti-VZV gE IgG for 2 doses of VNS vaccine compared to 2 doses of VV | At Day 133 (within 43 days post-dose 2)
  Concentrations of anti-VZV gE IgG are presented as GMC and expressed in mIU/mL for each group.

SECONDARY OUTCOMES:
Percentage of participants with seroresponse to anti-VZV gE IgG for VV-VNS group | At Day 133 (within 43 days post-dose 2)
  Seroresponse is defined as post-vaccination (Day 43 post Dose 2) anti-VZV gE IgG concentration >= 300 mIU/mL.
GMC of anti-VZV gE IgG for VV-VNS group | At Day 133 (within 43 days post-dose 2)
  Concentrations of anti-VZV gE IgG are presented as GMC and expressed in mIU/mL for each group.
Percentage of participants reporting each solicited administration site event | Day 1 (post-dose 1) to Day 4
  Solicited administration site events include injection site redness, pain and swelling.
Percentage of participants reporting each solicited administration site event | Day 91 (post-dose 2) to Day 94
  Solicited administration site events include injection site redness, pain and swelling.
Percentage of participants reporting each solicited systemic event | Day 1 (post-dose 1) to Day 15
  Solicited systemic events include drowsiness, loss of appetite and irritability.
Percentage of participants reporting each solicited systemic event | Day 91 (post-dose 2) to Day 105
  Solicited systemic events include drowsiness, loss of appetite and irritability.
Percentage of participants reporting each solicited systemic event in terms of fever | Day 1 (post-dose 1) to Day 22
  Fever is defined as temperature >=38.0 degrees Celsius (°C) by any route (the preferred location for measuring temperature is the axilla).
Percentage of participants reporting each solicited systemic event in terms of fever | Day 91 (post-dose 2) to Day 112
  Fever is defined as temperature >=38.0 degrees °C by any route (the preferred location for measuring temperature is the axilla).
Percentage of participants reporting each solicited administration site event | Day 1 (post-dose 1) to Day 43
  Solicited administration site include injection site varicella-like rash.
Percentage of participants reporting each solicited administration site event | Day 91 (post-dose 2) to Day 133
  Solicited administration site include injection site varicella-like rash.
Percentage of participants reporting each solicited systemic event | Day 1 (post-dose 1) to Day 43
  Solicited systemic events includes varicella-like rash (non-injection site), and general rash (not varicella-like).
Percentage of participants reporting each solicited systemic event | Day 91 (post-dose 2) to Day 133
  Solicited systemic events includes varicella-like rash (non-injection site), and general rash (not varicella-like).
Percentage of participants reporting unsolicited adverse events (AEs) | Day 1 (post-dose 1) to Day 43
  Unsolicited AEs include any AE reported in addition to solicited events during the study, or any "solicited" symptoms with onset outside of the specified period of follow-up for solicited symptoms, are assessed for each group after the administration of all vaccines.
Percentage of participants reporting unsolicited adverse events (AEs) | Day 91 (post-dose 2) to Day 133
  Unsolicited AEs include any AE reported in addition to solicited events during the study, or any "solicited" symptoms with onset outside of the specified period of follow-up for solicited symptoms, are assessed for each group after the administration of all vaccines.
Percentage of participants reporting medically attended AEs (MAAE) | Day 1 (post-dose 1) to Day 271 (study end)
  A MAAE is an AE for which the participant received medical attention including any symptom or illness requiring hospitalization, or an emergency room visit, or visit to/by a healthcare professional.
Percentage of participants reporting serious adverse events (SAEs) | Day 1 (post-dose 1) to Day 271 (study end)
  A SAE is an AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or other situations that are considered serious per medical or scientific judgment.

CONTACTS AND LOCATIONS:
Locations (3):
- Dominican Republic (3):
  - GSK Investigational Site, Salvaleón de Higüey, La Altagracia Province
  - GSK Investigational Site, Constanza
  - GSK Investigational Site, Santo Domingo Oeste

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf